CLINICAL TRIAL: NCT00702013
Title: Ontogenesis of the P-glycoprotein in Human Lymphocytes: Influence of the Human Immunodeficiency Virus (HIV) and Antiretroviral Therapeutics
Brief Title: Ontogenesis of the P-Glycoprotein in Human Lymphocytes Influence of HIV and Antiretroviral Therapeutics
Acronym: Onto-Pgp
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick Vacher, Department Clinical Research of Developpement
Other Study IDs: P070102
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infections
Keywords: P-glycoprotein; lymphocyte; HIV; children; ontogenesis; Ontogenesis P-gp in human lymphocytes; Study of the influence of HIV infection; Antiretroviral treatments on P-gp activity; Expression in human lymphocytes
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood sample for DNA extraction and genetic polymorphism of Mdr1
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- 1
- 2
- 3
- 4
- 5
- 6
- 7
- 8

SUMMARY:
The P-glycoprotein (P-gp) is a membranous transporter that modulates the intracellular concentrations of many drugs and plays thus a major role in the efficacy of the therapeutics that act within the lymphocytes, such as antiretroviral drugs. We aim at studying the evolution of this transporter's expression and activity on lymphocytes in relation with the human development from newborns to adults. We also aim at studying the influence of HIV and antiretroviral treatments on this transporter, especially anti-protease drugs, within the children population.

DETAILED DESCRIPTION:
Several groups of drugs involved in the treatment of major pathologies act within the lymphocyte, such as anticancer, immunosuppressive and antiretroviral drugs. These molecules depend on membranous transporters to get inside the lymphocyte and be effective. Among those transporters, the P-glycoprotein (P-gp) plays a major role, especially because of the variety of its substrates among therapeutic molecules. Its expression and activity are well known within the adult population, as well as its modulations mediated by certain groups of drugs, such as protease inhibitors in the treatment of HIV. Yet, there is very little data on children, even though they are exposed to the same therapeutic molecules as the adults. Therefore, we aim at studying the evolution of this transporter's expression and activity on the different lymphocyte populations, in relation to the human development from newborns to adults. We also aim at studying the influence of HIV and antiretroviral treatments on this transporter, especially anti-protease drugs, within the children population. P-gp activity is quantified by flow cytometry, through the efflux of a fluorescent substrate, in the presence or absence of a P-gp inhibitor. P-gp expression is measured on isolated motonucleus cells with the quantification of mRNA encoded for the transporter by RT-PCR (Reverse Transcription - Polymerase Chain Reaction). Patients of every age, from newborns to adults, are recruited within eight different age groups and three HIV status groups (HIV non infected, HIV infected untreated, HIV infected treated). The objective is to recruit ten patients in each age group for each HIV status. Blood samples are obtained from hospitalized children and adults with their consent. The patients will be recruited for one year. Our objective is to determine whether the P-gp expression and/or activity are influenced by age, HIV status and antiretroviral treatments, in order to prevent, depending on developmental stages, ineffectiveness or toxicity due to inadequate intracellular concentrations.

After the first evaluations, principal investigators decided to add one year more for three groups on eight.

For two groups of these three, genetic polymorphism of Mdr1 will be done.

ELIGIBILITY:
Inclusion Criteria:

* age, HIV status

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: HIV Patients children and adults and controls
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The activity and expression of P-glycoprotein at the time when the blood sample was taken. | immediately

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Tréluyer, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Necker Enfants Malades, Paris, France